CLINICAL TRIAL: NCT00820534
Title: A Randomised, Double-blind, Vehicle Controlled, Single Center, Parallel Group, Comparative Study of the Efficacy of Penciclovir 10mg/g (1%) Cream in Preventing the Appearance of Classical Lesion in Recurrent Cold Sore Sufferers
Brief Title: A Comparative Study of the Efficacy of Penciclovir 10mg/g (1%) Cream in Preventing the Appearance of Classical Lesion in Recurrent Cold Sore Sufferers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FPP4-DE-401
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2010-12

CONDITIONS: Cold Sore
Keywords: cold sore
MeSH Terms: conditions — Herpes Labialis | interventions — penciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Penciclovir (Experimental): Penciclovir
  Interventions: Drug: Penciclovir
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Penciclovir — Penciclovir every 2 hours during waking hours for 96 hours
  Arms: Penciclovir
Drug: Placebo — Placebo every 2 hous during waking hours for 96 hours
  Arms: Placebo

SUMMARY:
Comparison of the efficacy of penciclovir 10 mg/g (1%) cream with that of vehicle at 72 hours in preventing the appearance of classical lesions following prodromal symptoms (tingling or burning sensation) based on thermographic assessment among recurrent cold sore sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Be known to be a cold sore sufferer and presenting a prodromal stage with pain
* Sign the written informed consent form prior to enrolment in the trial;
* Be aged 18 to 75 years;

Exclusion Criteria:

* If female, are pregnant, planning pregnancy or lactating;
* Have a known hypersensitivity to penciclovir or any ingredients of the vehicle;
* Have already ongoing classical cold sore lesions at the baseline visit;
* Have taken any cold sore product, analgesic or NSAID in the 24 hours before the baseline visit;
* Have applied a cosmetic lip balm on their lips in the 12 hours before the baseline thermographic assessment;
* Are known to be immunosuppressed (acquired, congenital or therapeutic);
* Have been involved in any investigational protocol within the 30 days prior to the trial;
* Have evidence or history of drug or alcohol abuse;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lamey, Principal Investigator — Principal Investigator
Locations (1):
- Belfast Health and Social Care Trust, Royal Victoria Hospital, Belfast, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start : 30 dec 2008 Study end : 16 Nov 2009 Hospital out patient clinic
Pre-assignment Details: Cold Sore confirmed by local temperature measurement
Groups:
- Penciclovir: Penciclovir 10mg/g (1%) cream every 2 hours during waking hours for 96 hours
- Placebo: Placebo cream every 2 hours during waking hours for 96 hours
Period: Overall Study
Arm/Group | Penciclovir | Placebo
Started | 64 | 62
Completed | 64 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Penciclovir | Placebo | Total
Number analyzed (Participants) | 64 | 62 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 62 | 125
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 31.4 (11.3) | 31.8 (9.3) | 31.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United Kingdom | 64 | 62 | 126

OUTCOME MEASURES:

1. Primary Outcome: Clinical Assessment Performed by the Investigator and Skin Temperature at the Cold Sore.
Description: Number of participants where the classical cold sore lesion was prevented at 72 hours after first treatment application.Lesion defined as having been prevented if clinical assessment is prodrome, macule or healed and skin temperature of the cold sore is negative (temperature difference of less than 0.5°C between initial site of cold sore and opposite side).
Time Frame: 72 hours
Measure: Number; unit: participants
Arm/Group | Penciclovir | Placebo
Number analyzed (Participants) | 64 | 62
participants | 39 | 32

2. Secondary Outcome: Size of the Cold Sore
Description: The size of the cold sore was measured as follows : a standardized photograph was taken before treatment and compared to a photograph taken 72 hours after the first treatment application. The difference was calculated for each participant within each treatment arm.
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: square mm
Arm/Group | Penciclovir | Placebo
Number analyzed (Participants) | 64 | 62
square mm | 31.7 [20.8 to 42.6] | 32.7 [21.3 to 44.2]

ADVERSE EVENTS:
Arm/Group | Penciclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/62
Other Adverse Events (participants affected / at risk) | 0/64 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No